CLINICAL TRIAL: NCT03220074
Title: Efficacy and Tolerability of Linezolid for Treatment of Nontuberculous Mycobacterial Diseases
Brief Title: Linezolid for Treatment of Nontuberculous Mycobacterial Diseases
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mahidol University (Other)
Collaborators: Siam Pharmaceutical Ltd. (Unknown)
Responsible Party: Principal Investigator, Yupin Suputtamongkol, Professor, Mahidol University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Si268/2017
Record Dates: First submitted 2017-07-12; First posted 2017-07-18 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Non-tuberculous Mycobacterial Infections
MeSH Terms: interventions — Tablets

STUDY DESIGN:
Intervention Model Description: Open labelled study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment (Other): oral linezolid tablet 600 mg /day combine with either oral quinolone (ciprofloxacin or levofloxacin) or oral macrolide (azithromycin or clarithromycin)
  Interventions: Drug: Oral Tablet

INTERVENTIONS:
Drug: Oral Tablet — study drug given and monitored for efficacy and tolerability

SUMMARY:
A prospective open study to determine the efficacy and tolerability of oral linezolid 600mg./day for the treatment of 40 patients with nontuberculous mycobacterial diseases will be conducted at Siriraj Hospital, Mahidol University, Bangkok, Thailand.

DETAILED DESCRIPTION:
This will be an open label clinical study of oral linezolid combination with another oral antimycobacterial drug as the maintenance treatment of nontuberculous mycobacterial diseases in adult.

The eligible patients will be treated and monitored for the efficacy and safety every 6 weeks until 6 months then every 3 months for a total duration of 18 months.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of non-tuberculous mycobacterial (NTM) diseases
* Active or stable diseases receiving either parenteral or oral antimycobacterial treatment
* Require at least more than 6 months of treatment from enrollment

Exclusion Criteria:

* Stable NTM diseases with a plan to discontinue treatment within 3 months
* History of allergy to linezolid
* Hemoglobin < 7 g/dl) or total white blood count < 3,000 /cu.mm. or thrombocytopenia < 50,000 cells/cu.mm.
* Concomitant uses of serotoninergic drugs (SSRIs) or Monoamine oxidase inhibitor (MAOIs) within 30 days prior to enrollment
* Abnormal neurological findings such as numbness, abnormal vision etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-12-15 (Actual); Primary Completion 2021-06-15 (Actual); Study Completion 2022-06-15 (Actual)

PRIMARY OUTCOMES:
cure rate | 6 months
  no symptom and sign of active infection without drug treatment for at least 6 months

SECONDARY OUTCOMES:
rate of common adverse event (AE) | 18 months
  rate of common AE of linezolid such as thrombocytopenia, optic neuritis and rate of treatment withdrawal due to AEs

CONTACTS AND LOCATIONS:
Overall Officials: Yupin Suputtamongkol, MD, Principal Investigator — Mahidol University
Locations (1):
- Siriraj Hospital, Bangkoknoi, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Undecided